CLINICAL TRIAL: NCT06969950
Title: Evaluating an Evidence-Based Intervention for Physician Burnout
Brief Title: Evaluating an Intervention for Physician Burnout
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000677
Record Dates: First submitted 2025-03-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Physician Burnout
Keywords: burnout; physicians; app-based; smarthphone; mindfulness
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: One group will receive the intervention (audio-course) to listen during the study and the other group will have access to the audio-course at the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Early App-Delivered Mindfulness Training (MT). (Experimental): Participants will be asked to utilize the app designed to reduce burnout for 2 weeks
  Interventions: Other: App-Delivered Mindfulness Training (MT).
- Later App-Delivered Mindfulness Training (MT). (Other): Participants will receive the intervention after the three-month follow-up, not before.
  Interventions: Other: App-Delivered Mindfulness Training (MT).
- Experimental: Online Virtual Training (Experimental): A sub-group of participants will receive the virtual online training after three-month follow-up or directly after the app-based intervention.
  Interventions: Other: App-Delivered Mindfulness Training (MT).; Other: Online Virtual Training

INTERVENTIONS:
Other: App-Delivered Mindfulness Training (MT). — The program is delivered via a smartphone-based platform, which includes 7 mindfulness-based modules of about 15 minutes of brief didactic and experience-based for two weeks
Other: Online Virtual Training — A sub-group of 25 participants, either from the both intervention or control group, the will receive a virtual online training delivered via zoom calls. It is a group session program which includes 4 mindfulness-based sessions of about 60 minutes of brief didactic and experience-based for four weeks.
  Arms: Experimental: Online Virtual Training

SUMMARY:
The goals of this randomized controlled trial are 1) to test the efficacy of an app-based program in reducing physician burnout vs. no app (control) in 100 physicians; 2) to explore the role of an online live training to augment outcomes and develop an ongoing and sustainable support community with a subsample of physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Being a physician
2. Able to speak English because all study activities will be conducted in English.
3. 18+ years
4. Direct patient care

Exclusion Criteria:

1. If using psychotropic medication - not on a stable dosage at least 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Level of cynicism | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  Maslach Burnout Inventory (MBI) cynicism. The MBI is a validated 22-item self-report measure of risk of burnout. Items are rated on a 7-point Likert scale ranging from 0 (never) to 6 (every day). The investigators will use only one single-item measure of cynicism that was included from the Maslach Burnout Inventory (MBI)-based on the research of West et al., 2009.

SECONDARY OUTCOMES:
Level of emotional exhaustion | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  1.Maslach Burnout Inventory (MBI) emotional exhaustion. The MBI is a validated 22-item self-report measure of risk of burnout. Items are rated on a 7-point Likert scale ranging from 0 (never) to 6 (every day).
Level of anxiety | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  2.Generalized Anxiety Disorder 7-items (GAD-7). The GAD-7 is a validated 7-item measure of anxiety rated on a 4-point Likert scale ranging from 0 (Not at all sure) to 3 (Nearly every day).
Level of depression | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  Patient Health Questionnaire 2-item scale (PHQ-2). The PHQ-2 is a validated 2-item self-report measure of depression. Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
Level of intolerance of uncertainty | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  4.Intolerance of Uncertainty 12-item scale (IUS-12). The IUS-12 is a validated 12-item self-report measure of intolerance of uncertainty. Items are rated on a 5-point Likert scale ranging from 1 (not t all).
Level of self-compassion | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  5.Self-Compassion Scale. The SCS is a validated 12-item self-report measure of self-compassion on a 5-point Likert scale ranging from 1 (almost never) to 5 (always).

OTHER OUTCOMES:
Level of Work Engagement | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  1. Job Engagement Questionnaire (18 items). The Job Engagement questionnaire is a validated scale of the 18-item. This scale contains 18 items which are presented on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Level of patient-centered care | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  2. Nursing Workplace Satisfaction Questionnaire (NWSQ - 17). The NWSQ is a validated 17-item self-report measure of patient-centered care with items presented on a 5-point Likert scale ranging from 1 (fully disagree) to 5 (definitely disagree).
Level of organization civic behavior | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  3. Organizational Civic Behavior Scale (24 items). This questionnaire is a validated 24-item self-report measure of Organizational Civic Scale. Items are rated 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Level of physician well-being | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  4. Physician Well-Being Index (PWBI - 7 items). This questionnaire is a validated 7-item self-report measure of Physician Well-Being. Items are rated 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Level of loneliness | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  5. UCLA 3-Item Loneliness Scale (University California Los Angeles - 3 items). This questionnaire is a validated 3-item self-report measure of Loneliness. Items are rated 10-point Likert-type scale ranging from 1 (least lonely) to 10 (lost lonely).
Level of mindfulness practice | It will be collected 3 times, at baseline, 2 weeks after (post-app), three months later (follow-up). For the sub-group that will attend the online virtual training intervention, it will be collected after 4 months (post online training intervention).
  6. Mindful Practice Questionnaire (MIPR-Q - 28 items). This questionnaire is a validated 28-item self-report measure of Mindfulness practice. Items are rated 4-point Likert-type scale ranging from 1 (never/almost never) to 4 for (always/most always).
Elements learned | It will be collected one time, two weeks after the baseline (post-app). For the sub-group that will attend the online virtual training intervention, it will be collected a second time after 4 months (post online virtual training intervention).
  Open question regarding the elements learned with the app and virtual training sessions.
Facilitators | It will be collected one time, two weeks after the baseline (post-app). For the sub-group that will attend the online training intervention, it will be collected a second time after 4 months (post online training intervention).
  Open question regarding the facilitators encountered with the app and virtual training sessions.
Barriers | It will be collected one time, at two weeks after the baseline (post-app). For the sub-group that will attend the online virtual training, it will be collected a second time after 4 months (post online training intervention).
  Open question regarding the barriers encountered with the app and virtual training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Antico, PhD, Principal Investigator — Brown University; Joseph Casamassima, MSc, Study Chair — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No